CLINICAL TRIAL: NCT04234282
Title: Rate of Torque Development and Voluntary Quadriceps Activation in Patients With Knee Osteoarthritis: A Quantitative Analysis Before and After a Single Session of Manual Physical Therapy - A Randomized Controlled Trial
Brief Title: Rate of Torque Development and Voluntary Quadriceps Activation in Patients With Knee Osteoarthritis: A Quantitative Analysis Before and After a Single Session of Manual Physical Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jennifer Moreno Clinic (Other)
Responsible Party: Principal Investigator, MAJ Matthew Helton, Orthopedic and Manual Physical Therapy Fellow, Jennifer Moreno Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RTD_MVIC
Record Dates: First submitted 2019-11-13; First posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Knee Osteoarthritis; Knee Arthritis; Knee Pain Chronic; Knee Deformity; Knee Pain Swelling; Muscle Weakness; Muscle Weakness Condition; Power
MeSH Terms: conditions — Osteoarthritis, Knee; Muscle Weakness

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The patient will be randomly assigned using a random number generator to either the control or treatment group. The investigator and outcome assessor will not be present when the patient is receiving the control or treatment interventions. Pt will be instructed not to reveal which group they were assigned to when tested by the blinded assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group will receive a 30-minute class on knee osteoarthritis diagnosis, prognosis, various treatment options, and will conclude with a question and answer session. This will account for the 30 minute face to face time provided in the treatment group
- Manual Physical Therapy (Experimental): The treatment group will receive one 30-minute session of orthopedic manual physical therapy targeting the knee joint and soft tissues with complementary exercises targeted at their impairment. The manual therapy and exercises are tailored to the individual based on their limitations and restrictions.
  Interventions: Procedure: Manual Physical Therapy

INTERVENTIONS:
Procedure: Manual Physical Therapy — Orthopedic manual physical therapy targeting the knee joint and soft tissues with complementary exercises targeted at their impairment.
  Other Names: Joint Mobilization; Joint Manipulation
  Arms: Manual Physical Therapy

SUMMARY:
This is a randomized control trial to determine if there is a measurable change in voluntary quadriceps activation, RTD, pain, and function before and after a single session of manual physical therapy.

The researchers will utilize a sample of convenience with consecutive sampling at the Brooke Army Medical Center physical therapy clinic for patients referred for knee osteoarthritis.

As is standard of care, patients will be provided a medical intake form and a clinical outcome measure commensurate with their primary anatomic region for which they are seeking physical therapy (i.e.: Lower Extremity Functional Scale for hip, knee, or ankle pain). If patients choose to partake in the study, they will complete the consent form and the initial physical therapy evaluation will be conducted. They will then be provided an appointment for data collection at the Army-Baylor Center for Rehabilitation Research biomechanics lab at the Army Medical Department Center and School.

The treatment group will receive one 30-minute session of orthopedic manual physical therapy targeting the knee joint and soft tissues with complementary exercises targeted at their impairment.

The control group will receive a 30-minute class on knee OA diagnosis, prognosis, various treatment options, and will conclude with a question and answer with the researcher. Both groups will receive their intervention from a board-certified physical therapist in the Army-Baylor Orthopedic Manual Therapy Fellowship program.

At the conclusion of formal testing, the patient will be provided standard physical therapy care as deemed appropriate by their evaluating physical therapist. Thus, all subjects, regardless of their assigned group, will receive the same standard of care for their knee pain.

DETAILED DESCRIPTION:
By participating in this study, it will not alter the standard of care provided during the course of the patient's rehabilitation in physical therapy. During the initial physical therapy evaluation, a member of the research team will determine if the patient would like to participate in the study and if they choose to do so they will then be consented. Based on the clinical presentation the standard evaluation will determine the primary limitations of the knee joint and surrounding soft tissue structures and outline the best course of manual physical therapy intervention deemed appropriate.

Should the patient choose to participate, they will then complete a pre-test maximal isometric contraction in the knee extension machine in the physical therapy clinic; this is an exercise device commonly used to strengthen the quadriceps muscles for patients with various types of lower extremity pathology. Patients will be monitored for any changes in pain during this screening pre-test in accordance with the Physical Therapy service standard operating procedures; those whom pain increases more than 3/10 points on the numeric pain rating scale from baseline will be excluded from this study and will be counted as screen failures; all others will be included in the study. The patient will then be provided an appointment slip to meet the research team at the Army-Baylor Center for Rehabilitation Research Biomechanics Lab at the Army Medical Department Center and School where all formal testing for this study will take place. All laboratory data will be collected for the bilateral lower extremities.

When the subject reports to the lab the following sequence will occur. They will be provided with an intake form to collect all baseline data, Western Ontario and McMaster Universities Osteoarthritis Index, and numeric pain rating score. Pain scores will be elicited throughout the testing procedures to ensure patient safety and comfort per the PT service pain assessment standard operating procedures. Pain pressure threshold will be obtained using a handheld algometer as an adjunct to the numeric pain rating scale to better quantify their pain levels. Pain pressure threshold measures will be collected bilaterally over the Tibialis Anterior muscle belly approximately 2.5cm lateral and 5cm inferior to the tibial tubercle. A Timed up and Go test will then be administered using an accelerometer worn by the patient around the waist and bilaterally on the dorsum of the foot to quantify the velocity in which they complete the test among the various phases (sit/stand, walking, turning). This will be followed by the first isometric testing session to determine the baseline voluntary quadriceps activation and rate of torque development.

Subjects will undergo assessment of neuromuscular function using a combination of voluntary and evoked contractions. All test procedures will be performed on the unaffected limb first, followed by the affected limb. Electrically-evoked contractile properties will be tested first, followed by volitional strength, voluntary activation, then rate of torque development.

Subjects will be seated on the chair for the HUMAC NORM testing and rehabilitation system with the hips and knees flexed to 85 degrees and 60 degrees, respectively. A shin attachment from the dynamometer will be secured around the subjects' lower leg so that the distal end of the pad is approximately 5 cm proximal to the distal end of the tibia anteriorly.

Two-inch by four-inch self-adhesive muscle stimulation electrodes will be applied over the muscle bellies of the distal vastus medialis and proximal vastus lateralis. Subjects will then undergo evoked twitch contractions starting at 50mA (400 V, 1000 µsec pulse width) using a constant current muscle and nerve stimulator (Digitimer Ltd., Model DS7R, Hertfordshire, England) while sitting at rest. This process will continue until the evoked torque reaches a plateau, at which point it will be terminated. The purpose of this testing is to determine the lowest intensity of current necessary to evoke maximal quadriceps torque for each subject. The amount of current necessary to achieve peak evoked twitch torque will be used for all future evoked contractions. After this, muscle speed properties will be assessed using 3 maximal twitches, followed by 3 maximal doublets at 100 Hz, all 10 seconds apart from each other. This will be done for a total of 6 evoked contractions. The purpose of this is to obtain information related to the peripheral speed properties of the muscle (e.g., rates of rise and relaxation for torque).

Maximum volitional isometric contraction testing will be assessed next. Strength testing will begin by having subjects perform 3 sub-maximal (50%, 75%, 90% maximum effort) isometric knee extension contractions to familiarize themselves. After familiarization, subjects will perform at least 2 maximal voluntary isometric contractions of the quadriceps muscles to determine the peak voluntary knee extensor force each subject can generate. For reliability, the researchers will require two contractions that produce similar values of torque (defined as no more than 5% difference between trials). After peak torque has been reliably identified, quadriceps activation will be tested with the interpolated doublet technique (IDT).[30] This test includes at least two five second maximal voluntary isometric contractions during which a doublet at the stimulus intensity determined in step one is introduced when the torque produced by the subject reaches a threshold determined during maximal voluntary isometric contraction testing. A second stimulus of equal intensity is delivered shortly after the subject returns to rest after each trial in order to assess the muscle in its potentiated state. Two minutes rest will be provided between each of the trials. To produce inter-trial reliability similar to strength testing, the researchers will require two contractions that produce similar values of voluntary activation (defined as no more than 5% difference in voluntary activation between trials).

Rate of torque development will be measured after completion of maximal voluntary isometric contraction trials. A total of five valid repetitions will be completed lasting approximately one second in duration for each contraction. In order to count as a valid trial, the magnitude of torque attained during these brief contractions must exceed 75% of maximal voluntary isometric contraction. A rest period of 30 seconds between contractions will be given in order to allow for adequate rest. An enthusiastic and loud verbal cue will be provided for each contraction. Instructions to "kick as fast and as hard as possible" will be utilized as verbal cues have been reported to impact the type of motion the patient conducts. Visual feedback and loud verbal encouragement will be used to elicit the greatest amount of muscle activation possible.

Treatment will be initiated within ten minutes of completing the first isometric trial within the Army-Baylor Center for Rehabilitation Research. The researchers will utilize a pragmatic manual physical therapy approach that is customized to each subject. This approach will use targeted manual therapy techniques for the knee joint and soft tissues with complimentary therapeutic exercises to augment the movement impairment identified. All treatment will be performed by a board-certified physical therapist with advanced manual physical therapy fellowship training. The treatment provided will be evidenced-based and is standard care for a manual physical therapy trained provider. The timing of the treatment session is congruent with what is commonly observed in a physical therapy clinic and will last approximately 30 minutes in duration.

The control group will receive the same amount of face-to-face time with a physical therapist. The intervention will include a 30-minute educational class on knee osteoarthritis which will cover various topics to include a brief description of the pathophysiology, diagnosis, prognosis, and different treatment options available in addition to rehabilitation. The researchers will provide handouts on general exercise and joint sparing activities and conclude the brief with a question and answer session.

For post-treatment data collection, each subject will undergo testing for maximal voluntary isometric contraction, voluntary activation, and rate of torque development in the same manner as described above. For voluntary activation testing, the same stimulus intensity determined during pre-treatment data collection will be used. In addition, subjects will not require post-treatment assessment of the contractile properties of their quadriceps muscle group. The reason for not repeating this assessment is because electrically-evoked contractile properties quantify only peripheral physiologic properties of muscle and this study's intent is to measure changes attributed to central drive (i.e. changes within the motor cortex and/or spinal cord).

Immediately following the 30-minute treatment session, subjects will repeat the timed up and go test and rate their pain via the numeric pain rating scale. Immediately following this, the subject will undergo maximal voluntary isometric contraction testing, voluntary activation, and rate of torque development testing in the same manner previously described. The same stimulator settings used during the pre-test will be used for the post-test. At the conclusion of data collection, the researchers will ensure the patient has a follow-up appointment scheduled at the Brooke Army Medical Center physical therapy clinic for the initiation of their formal rehabilitation, thus ensuring that all subjects receive the standard of care for their knee pain. As all data will be collected on a single day in one session no email or phone calls will be required at the completion of the lab testing.

ELIGIBILITY:
Inclusion Criteria:

* Age range including 50-70 years old
* Diagnosis of clinical and radiographic knee osteoarthritis (Altman's Criteria: knee pain, osteophytes and one of the following: crepitus with active motion, morning stiffness less than or equal to 30 minutes, bony enlargement)
* Grade 2-4 Kellgren Lawrence radiographic knee osteoarthritis

Able to tolerate maximal quadriceps isometric quadriceps contraction with the knee flexed to 60 degrees without pain increasing more than 3/10 points on the Numeric Pain rating scale

5

* English proficiency and cognition to understand explanations of research purpose and procedures
* Tricare beneficiary

Exclusion Criteria:

* Knee pain referred from another anatomic region
* Cardiovascular disease (limited to uncontrolled hypertension/arrhythmias as well as a pacemaker
* Rheumatoid arthritis
* Active cancer
* BMI > 35
* Intra-articular knee injection within the previous 3 months
* Traumatic knee injury or surgery in past 12months
* Total knee or hip arthroplasty
* Gait is limited to a greater extent by conditions other than knee osteoarthritis
* Any condition that would contraindicate manual therapy or exercise
* Medical "red flags" of a potentially serious condition including cauda equina syndrome, major or rapidly progressing neurological deficit, fracture, active infection, or systemic disease
* Known current pregnancy or history of pregnancy in the last 6 months
* Separating from the military in the next 2 months, pending litigation, or pending medical board

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Rate of Torque Development | 3 hours
  The between-session reliability for quadriceps peak torque (ICC2,3 = 0.98) has been shown to be optimized by performing five repetitions and using the average of the three repetitions with the highest isometric peak torque with a 30 second rest period between contractions. The minimal detectable change for healthy controls is reported as 265.4 Nm/s with a standard deviation of 112.8 Nm/s.[29]
Voluntary Quadriceps Activation | 3 hours
  This variable will be calculated utilizing the interpolated twitch technique by superimposing an electrical stimulus to quadriceps maximum volitional isometric contraction and using the same stimulus applied at rest. Interpolated twitch technique is an accurate method to calculate voluntary quadriceps activation.[30, 35]

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | 3 hours
  The Numeric Pain Rating Scale is a self-reported 11-point scale from 0-10 for pain intensity, which has been shown to be sensitive to change and has been shown to be valid and reliable for patients with chronic pain. The minimally clinically important difference has been reported as 2 on this scale.
Timed Up and Go Test | 3 hours
  The Timed Up and Go test has been shown to be sensitive to small changes in functional status and may be a good indicator to measure the progress of rehabilitation interventions. The decrease in time to conduct the Timed Up and Go Test by as little as .8 seconds has been associated with improved Global Rating of Change scores of +5. This measure has been shown to be reliable and is a good indicator of physical mobility in older frail adults. [33]

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S Helton, DPT, Principal Investigator — Orthopedic PT Fellow
Locations (1):
- Jennifer Moreno Clinic, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patients' confidentiality will be protected in the data collection process. All paper copies of study files will be stored in a locked cabinet in the Manual Physical Therapy Fellowship classroom inside the Moreno Clinic. Consent forms that identify the patient by name will be stored in a locked cabinet separately from the remainder of the outcome instruments. The data file linking the names and code numbers will be accessible only to the Principal Investigator, and data from each individual will be entered into a computer file by this code number on a password protected/ common access card enabled computer.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The informed consent document will be kept for 3 years.
Access Criteria: Orthopedic Manual Physical Therapy Fellowship Director or Fellow

REFERENCES:
- [Background] 1. Showery, J.E., et al., The rising incidence of degenerative and posttraumatic osteoarthritis of the knee in the United States military. 2016. 31(10): p. 2108-2114. 2. Armed, F.H.S.B.J.M., Absolute and relative morbidity burdens attributable to various illnesses and injuries, non-service member beneficiaries of the Military Health System, 2017. 2018. 25(5): p. 32. 3. Zhang, Y. and J.M.J.C.i.g.m. Jordan, Epidemiology of osteoarthritis. 2010. 26(3): p. 355-369. 4. Milley, M.A.J.U.S.A., 39th Chief of Staff initial message to the army. 2015. 5. Anwer, S., et al., Effects of orthopaedic manual therapy in knee osteoarthritis: a systematic review and meta-analysis. 2018.
- [Background] 11. Fitzgerald, G.K., et al., Quadriceps activation failure as a moderator of the relationship between quadriceps strength and physical function in individuals with knee osteoarthritis. Arthritis Rheum, 2004. 51(1): p. 40-8. 12. Petterson, S.C., et al., Mechanisms undlerlying quadriceps weakness in knee osteoarthritis. 2008. 40(3): p. 422. 13. Rice, D.A., et al., Mechanisms of quadriceps muscle weakness in knee joint osteoarthritis: the effects of prolonged vibration on torque and muscle activation in osteoarthritic and healthy control subjects. 2011. 13(5): p. R151. 14. Rice, D.A. and P.J. McNair. Quadriceps arthrogenic muscle inhibition: neural mechanisms and treatment perspectives. in Seminars in arthritis and rheumatism. 2010. Elsevier. 15. Maffiuletti, N.A., et al., Rate of force development: physiological and methodological considerations. 2016. 116(6): p. 1091-1116.
- [Background] 21. Deyle, G.D., et al., Knee OA: which patients are unlikely to benefit from manual PT and exercise? 2012. 61(1): p. E1-8. 22. Deyle, G.D., et al., Effectiveness of manual physical therapy and exercise in osteoarthritis of the knee: a randomized, controlled trial. 2000. 132(3): p. 173-181. 23. Taylor, A.L., et al., Knee extension and stiffness in osteoarthritic and normal knees: a videofluoroscopic analysis of the effect of a single session of manual therapy. 2014. 44(4): p. 273-282. 24. Maitland, G.D., et al., Maitland's vertebral manipulation. Vol. 1. 2005: Elsevier Butterworth-Heinemann Philadelphia, PA. 25. Grindstaff, T.L., et al., Effects of lumbopelvic joint manipulation on quadriceps activation and strength in healthy individuals. Man Ther, 2009. 14(4): p. 415-20.
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] 6. Øiestad, B., et al., Knee extensor muscle weakness is a risk factor for development of knee osteoarthritis. A systematic review and meta-analysis. 2015. 23(2): p. 171-177. 7. Felson, D.T., et al., The prevalence of knee osteoarthritis in the elderly. The Framingham Osteoarthritis Study. 1987. 30(8): p. 914-918. 8. Vina, E.R. and C.K. Kwoh, Epidemiology of osteoarthritis: literature update. Curr Opin Rheumatol, 2018. 30(2): p. 160-167. 9. Guccione, A.A., et al., The effects of specific medical conditions on the functional limitations of elders in the Framingham Study. Am J Public Health, 1994. 84(3): p. 351-8. 10. Slemenda, C., et al., Quadriceps weakness and osteoarthritis of the knee. Ann Intern Med, 1997. 127(2): p. 97-104.
- [Background] 16. Cobian, D.G., et al., Knee Extensor Rate of Torque Development Before and After Arthroscopic Partial Meniscectomy, With Analysis of Neuromuscular Mechanisms. 2017. 47(12): p. 945-956. 17. Folland, J., et al., Human capacity for explosive force production: neural and contractile determinants. 2014. 24(6): p. 894-906. 18. Jevsevar, D.S.J.J.-J.o.t.A.A.o.O.S., Treatment of osteoarthritis of the knee: evidence-based guideline. 2013. 21(9): p. 571-576. 19. Nussmeier, N.A., et al., Complications of the COX-2 inhibitors parecoxib and valdecoxib after cardiac surgery. 2005. 352(11): p. 1081-1091. 20. SooHoo, N.F., et al., Factors predicting complication rates following total knee replacement. 2006. 88(3): p. 480-485.
- [Background] 26. Suter, E., et al., Conservative lower back treatment reduces inhibition in knee-extensor muscles: a randomized controlled trial. J Manipulative Physiol Ther, 2000. 23(2): p. 76-80. 27. Yerys S, M.H., Byrd C, Pennachio J, Cinkay J, Effect of mobilization of the anterior hip capsule on gluteus maximus strength. Journal of Manual & Manipulative Therapy, 2002(10): p. 218-224 . 28. Makofsky H, P.S., Abbruzzese J, Aridas C, Camp M, Drakes J, Franco C, Sileo R, Immediate Effect of Grade IV Inferior Hip Joint Mobilization on Hip Abductor Torque: A Pilot Study. Journal of Manual & Manipulative Therapy, 2007. 15: p. 103-111. 29. Grindstaff, T.L., et al., Optimizing Between-Session Reliability for Quadriceps Peak Torque and Rate of Torque Development Measures. 2018. 30. Krishnan, C. and G.N. Williams, Quantification method affects estimates of voluntary quadriceps activation. Muscle Nerve, 2010. 41(6): p. 868-74.
- [Background] Kean CO, Birmingham TB, Garland SJ, Bryant DM, Giffin JR. Minimal detectable change in quadriceps strength and voluntary muscle activation in patients with knee osteoarthritis. Arch Phys Med Rehabil. 2010 Sep;91(9):1447-51. doi: 10.1016/j.apmr.2010.06.002. PMID 20801266
- [Background] 33. Podsiadlo, D. and S.J.J.o.t.A.g.S. Richardson, The timed "Up & Go": a test of basic functional mobility for frail elderly persons. 1991. 39(2): p. 142-148. 34. Bennell, K., et al., Measures of physical performance assessments: Self Paced Walk Test (SPWT), Stair Climb Test (SCT), Six Minute Walk Test (6MWT), Chair Stand Test (CST), Timed Up & Go (TUG), Sock Test, Lift and Carry Test (LCT), and Car Task. 2011. 63(S11): p. S350-S370. 35. Zarkou, A., et al., Comparison of techniques to determine human skeletal muscle voluntary activation. J Electromyogr Kinesiol, 2017. 36: p. 8-15.